CLINICAL TRIAL: NCT03571087
Title: A Multi Center, Randomized, Double-blind, Parallel, Factorial Design, Therapeutic Phase III Study to Evaluate the Efficacy and Safety of Combination of Rosuvastatin and Ezetimibe in Patients With Primary Hypercholesterolemia
Brief Title: Efficacy and Safety of Combination of Rosuvastatin and Ezetimibe in Patients With Primary Hypercholesterolemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hanlim Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HL_HL140_301
Record Dates: First submitted 2018-06-17; First posted 2018-06-27 (Actual); Last update posted 2018-08-14 (Actual); Status verified 2018-06

CONDITIONS: Primary Hypercholesterolemia
MeSH Terms: interventions — Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- HL140 5/10 (Experimental): Treatment(W0~W8), Extension(W9~W20): : 6Tab./q.d. HL140 5/10(Rosuvastatin5mg/Ezetimibe10mg)
  Interventions: Drug: HL140 5/10
- HL140 10/10 (Experimental): Treatment(W0~W8), Extension(W9~W20): : 6Tab./q.d. HL140 10/10(Rosuvastatin10mg/Ezetimibe10mg)
  Interventions: Drug: HL140 10/10
- HL140 20/10 (Experimental): Treatment(W0~W8), Extension(W9~W20): : 6Tab./q.d. HL140 20/10(Rosuvastatin20mg/Ezetimibe10mg)
  Interventions: Drug: HL140 20/10
- Rosuvastatin 5mg → HL140 5/10 (Experimental): 1. Treatment(W0~W8): 6Tab./q.d. Rosuvastatin 5mg
  2. Extension period(W9~W20): 6Tab./q.d. HL140 5/10(Rosuvastatin5mg/Ezetimibe10mg)
  Interventions: Drug: Rosuvastatin 5mg → HL140 5/10
- Rosuvastatin 10mg → HL140 10/10 (Experimental): 1. Treatment(W0~W8): 6Tab./q.d. Rosuvastatin 10mg
  2. Extension period(W9~W20): 6Tab./q.d. HL140 10/10(Rosuvastatin10mg/Ezetimibe10mg)
  Interventions: Drug: Rosuvastatin 10mg → HL140 10/10
- Rosuvastatin 20mg → HL140 20/10 (Experimental): 1. Treatment(W0~W8): 6Tab./q.d. Rosuvastatin 20mg
  2. Extension period(W9~W20): 6Tab./q.d. HL140 20/10(Rosuvastatin20mg/Ezetimibe10mg)
  Interventions: Drug: Rosuvastatin 20mg → HL140 20/10

INTERVENTIONS:
Drug: HL140 5/10 — 1) Treatment(W0~W8), Extension(W9~W20): 6Tab./q.d. HL140 5/10(Rosuvastatin5mg/Ezetimibe10mg) : ●♤♡□△◇
  ●: HL140 5/10mg, ♤: HL140 10/10mg placebo, ♡: HL140 20/10mg placebo, □: Crestor Tab.5mg placebo, △: Crestor Tab. 10mg placebo, ◇: Crestor Tab. 20mg placebo
  Arms: HL140 5/10
Drug: HL140 10/10 — 1) Treatment(W0~W8), Extension(W9~W20): 6Tab./q.d. HL140 10/10(Rosuvastatin10mg/Ezetimibe10mg) : ○♠♡□△◇
  ○: HL140 5/10mg placebo, ♠: HL140 10/10mg, ♡: HL140 20/10mg placebo, □: Crestor Tab. 5mg placebo, △: Crestor Tab. 10mg placebo, ◇: Crestor Tab. 20mg placebo
  Arms: HL140 10/10
Drug: HL140 20/10 — 1) Treatment(W0~W8), Extension(W9~W20): 6Tab./q.d. HL140 20/10(Rosuvastatin20mg/Ezetimibe10mg) : ○♤♥□△◇
  ○: HL140 5/10mg placebo, ♤: HL140 10/10mg placebo, ♥: HL140 20/10mg, □: Crestor Tab. 5mg placebo, △: Crestor Tab. 10mg placebo, ◇: Crestor Tab. 20mg placebo
  Arms: HL140 20/10
Drug: Rosuvastatin 5mg → HL140 5/10 — 1. Treatment(W0~W8): 6Tab./q.d. Rosuvastatin 5mg : ○♤♡■△◇
     ○: HL140 5/10mg placebo, ♤: HL140 10/10mg placebo,♡: HL140 20/10mg placebo, ■: Crestor Tab. 5mg, △: Crestor Tab. 10mg placebo, ◇: Crestor Tab. 20mg placebo
  2. Extension period(W9~W20): 6Tab./q.d. HL1405/10(Rosuvastatin5mg/Ezetimibe10mg) : ●♤♡□△◇
     * HL140 5/10mg, ♤: HL140 10/10mg placebo, ♡: HL140 20/10mg placebo, □: Crestor Tab. 5mg placebo, △: Crestor Tab. 10mg placebo, ◇: Crestor Tab. 20mg placebo
  Arms: Rosuvastatin 5mg → HL140 5/10
Drug: Rosuvastatin 10mg → HL140 10/10 — 1. Treatment(W0~W8): 6Tab./q.d. Rosuvastatin 10mg : ○♤♡□▲◇
     ○: HL140 5/10mg placebo, ♤: HL140 10/10mg placebo, ♡: HL140 20/10mg placebo, □: Crestor Tab. 5mg placebo, ▲: Crestor Tab. 10mg, ◇: Crestor Tab. 20mg placebo
  2. Extension period(W9~W20): 6Tab./q.d. HL140 10/10(Rosuvastatin10mg/Ezetimibe10mg) : ○♠♡□△◇
     * HL140 5/10mg placebo, ♠: HL140 10/10mg, ♡: HL140 20/10mg placebo, □: Crestor Tab. 5mg placebo, △: Crestor Tab. 10mg placebo, ◇: Crestor Tab. 20mg placebo
  Arms: Rosuvastatin 10mg → HL140 10/10
Drug: Rosuvastatin 20mg → HL140 20/10 — 1. Treatment(W0~W8): 6Tab./q.d.Rosuvastatin 20mg : ○♤♡□△◆
     ○: HL140 5/10mg placebo, ♤: HL140 10/10mg placebo, ♡: HL140 20/10mg placebo, □: Crestor Tab. 5mg placebo, △: Crestor Tab. 10mg placebo, ◆: Crestor Tab. 20mg
  2. Extension period(W9~W20): 6Tab./q.d. HL140 20/10(Rosuvastatin20mg/Ezetimibe10mg) : ○♤♥□△◇ ○: HL140 5/10mg placebo, ♤: HL140 10/10mg placebo, ♥: HL140 20/10mg, □: Crestor Tab. 5mg placebo, △: Crestor Tab. 10mg placebo, ◇: Crestor Tab. 20mg placebo
  Arms: Rosuvastatin 20mg → HL140 20/10

SUMMARY:
The purpose of this study is to evaluate efficacy and safety of HL140 in patients with primary hypercholesterolemia.

DETAILED DESCRIPTION:
The purpose of this study is to demonstrate that the efficacy of combination drug of rosuvastatin/ezetimibe is superior to single rosuvastatin drug and to confirm the safety of combination drug of rosuvastatin/ezetimibe

ELIGIBILITY:
Inclusion Criteria:

* Aged over 19 years
* Signed informed consent form
* At visit 1 and visit 2, LDL-Cholesterol ≤ 250mg/dL and Triglyceride ≤ 400mg/dL

Exclusion Criteria:

* At visit 1, BMI ≥ 30kg/㎡
* Has a history of myopathy or rhabdomyolysis cased by statin treatment, hereditary myopathy or family history and hypersensitivity to statin(HMG-CoA reductase inhibitor) and component of ezetimibe
* Has a Severe renal disorder(Ccr <30mL/min) or nephrotic syndrome
* Creatine Kinase > 5 x upper limit of normal
* ALT or AST > 3 x upper limit of normal
* Has a activity/chronic hepatic disease or HIV-positive
* Has a endocrine or metabolic diseases known to affect the serum phospholipid or protein

  * Uncontrolled diabetes mellitus(HbA1c ≥9%)
  * Hypothyroidism (TSH > 1.5 x upper limit of normal rate at the screening )
* Uncontrolled hypertension (SBP ≥180mmHg or DBP ≥110mmHg)
* Has a acute arteriopathy(history of unstable angina, cardiac infarction, transient ischemic stroke, cerebrovascular disease, coronary artery bypass, coronary intervention within 12 weeks prior to screening)
* Severe heart failure (NYHA Class III or IV)
* Has a drug absorption disorder by gastrointestinal surgery or gastrointestinal disorder
* History of malignant tumor including myelogenous and lymphoma within 5 years (Participation is possible, if the tumor has not recurred for more than 5 years)
* Subject with genetic deficiency such as galactose intolerance, Lapp lactose deficiency or glucose-galactose malabsorption
* Female subjects of childbearing potential who disagree with the contraceptive methods(surgical sterilization, intrauterine device or condoms)
* Pregnant or breast-feeding
* Patients who have a drug or alcohol abuse or are being treated for psychological disorder
* Patients who were treated with other investigational drug within 12 weeks prior to screening
* Other patients who are inappropriate to participate in the study considered by the investigator or other study staffs

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 374 (Actual)
Dates: Start 2014-09; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Percentage change in LDL-Cholesterol from baseline | Week 8
  Percentage change(%) in LDL-Cholesterol from baseline at week 8

SECONDARY OUTCOMES:
Percentage change in LDL-Cholesterol from baseline | Week 4
  Percentage change(%) in LDL-Cholesterol from baseline at week 4
Percentage change in TG from baseline | Week 4, Week 8
  Percentage change(%) in TG from baseline at week 4 and week 8
Percentage change in TC from baseline | Week 4, Week 8
  Percentage change(%) in TC from baseline at week 4 and week 8
Percentage of change in non-HDL-Cholesterol | Week 4, Week 8
  Percentage change(%) in non-HDL-Cholesterol from baseline at week 4 and week 8
Percentage of change in HDL-Cholesterol | Week 4, Week 8
  Percentage change(%) in HDL-Cholesterol from baseline at week 4 and week 8
Percentage of change weeks in Apo A-I | Week 4, Week 8
  Percentage change(%) in Apo A-I from baseline at week 4 and week 8
Percentage of change in Apo B | Week 4, Week 8
  Percentage change(%) in Apo B from baseline at week 4 and week 8
Percentage of change in Lipoprotein(a) | Week 4, Week 8
  Percentage change(%) in Lipoprotein(a) from baseline at week 4 and week 8
The rate of change in hs-CRP | Week 4, Week 8
  Percentage change(%) in hs-CRP from baseline at week 4 and week 8
Percentage of patients reached treatment goals according to NCEP ATP III Guideline | Week 4, Week 8
  Percentage(%) of patients reached treatment goal, by NCEP ATP III guideline, at week 4 and week 8

CONTACTS AND LOCATIONS:
Overall Officials: Kisik Kim, Study Chair — The Catholic University of Korea, Dagu St. Mary's Hospital